CLINICAL TRIAL: NCT05331222
Title: Proof-of-Concept Interventional Study With a Nasal Spray of JT-1 in Patients With Chronic Rhinitis or Chronic Sinusitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: regulatory issues
Sponsor: Jantar GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2021-00564
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Chronic Rhinitis; Chronic Sinus Congestion
Keywords: rhinitis, sinusitis, rhinosinusitis
MeSH Terms: conditions — Rhinitis; Sinusitis; Rhinosinusitis

STUDY DESIGN:
Intervention Model Description: Single-arm proof-of-concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jantar-1 (JT-1), 7% (w/w) aqueous solution (Experimental): Dosing regimen: ad libitum between at least 2 doses, in the morning and in the evening, and at most 10 doses per day. A dose corresponds to two strokes of 100ul each per nostril.
  Interventions: Drug: JT-1

INTERVENTIONS:
Drug: JT-1 — JT-1 is a physiological salt with recently detected pharmacological properties that warrant testing for its therapeutic potential in chronic rhinitis and chronic sinusitis.

SUMMARY:
Proof-of-concept study with a novel nasal spray in chronic rhinitis or chronic sinusitis. The study will involve 25 patients completing the study for a per protocol analysis.

DETAILED DESCRIPTION:
Visit 1 (Day 0): Screening visit. Assessment of outcome measures

Visit 2 (Day 7): Enrollment visit after a 1-week wash-out period. Enrolled to the Study are only patients who show a severe enough and stable disease (SNOT score >20 and change of SNOT score <15% compared to Visit 1, respectively).

Visit 3 (Day 21): Assessment of outcome measures after 2-week treatment phase

Visit 4 (Day 49): Follow-up visit

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed chronic allergic rhinitis or chronic sinusitis with no or a mild status of nasal polyp activity
* Disease lasting 12 weeks or longer
* Patients with moderate or severe symptoms (SNOT-22 score >20)
* Male or female at least 18 years old
* Females in childbearing age are requested to make a pregnancy test and to confirm in writing to take contraceptive measures until Follow-up Visit (Day 49).
* Patient understands German

Exclusion Criteria:

* Severely purulent forms of sinusitis
* History of medication during the last four weeks

  * not allowed: antibiotics, systemic or topical steroids
  * allowed: nasal saline spray or irrigation, analgesics, decongestants, antihistamines
* Patient has a status of moderate or severe polyp activity in the nose
* Patient had sinus surgery in the past 6 months
* Patient needs O2 substitution
* Patient has cystic fibrosis
* Patient has primary ciliary dyskinesia
* Patient is demented or otherwise incapable of judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Change of Sino-Nasal Outcome Test (SNOT) score from baseline | Baseline (enrollment visit) and after 2-week treatment phase
  Questionnaire of 22 questions on the subjective clinical symptoms of chronic rhinitis and chronic sinusitis, score between 0 (no symptoms) and 120 (worst possible disease)

SECONDARY OUTCOMES:
Change of Peak Nasal Inspiratory Flow (PNIF) from baseline | Baseline (enrollment visit) and after 2-week treatment phase
  The PNIF meter measures the nasal airway patency in L/min.
Change of Smell Diskettes Olfactory Test from baseline | Baseline (enrollment visit) and after 2-week treatment phase
  Standardized 8-item odor (forced multiple choice) identification test (score of 0 to 8 correct answers)
Change of Visual Analog Scale (VAS) of Headache Intensity | Baseline (enrollment visit) and after 2-week treatment phase
  VAS is a method to measure the symptom severity. Patients mark a spot on a 100mm long line between no pain (left end) and worst possible pain (right end) which corresponds to their current pain level. The distance between the left end and the mark measures the subjective severity of pain. Minimum value: 0; maximum value: 100. A lower score after treatment compared to baseline means improved outcome.
Change of Visual Analog Scale (VAS) of Nasal Discomfort | Baseline (enrollment visit) and after 2-week treatment phase
  VAS is a method to measure the symptom severity. Patients mark a spot on a 100mm long line between no discomfort (left end) and worst possible discomfort (right end) which corresponds to their current level of discomfort. The distance between the left end and the mark measures the subjective severity of nasal discomfort. Minimum value: 0; maximum value: 100. A lower score after treatment compared to baseline means improved outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Rudolf Briner, KD MD, Principal Investigator — ORL-Center, Clinic Hirslanden, Zurich, Switzerland
Locations (1):
- Clinic Hirslanden, ORL-Center, Zurich, Canton of Zurich, Switzerland